CLINICAL TRIAL: NCT00759993
Title: A 6 Week, Blinded, Randomized, Controlled Pilot Study to Evaluate the Safety and Efficacy of Chromium Piccolinate in the Prevention of Weight Gain Induced by Serotonergic Medications Initiated on Psychiatric Inpatient Units.
Brief Title: Chromium Piccolinate in the Prevention of Weight Gain Induced by Serotonergic Medications Initiated on Psychiatric Inpatient Units.
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: inability to recruit and retain
Sponsor: State University of New York - Upstate Medical University (Other)
Collaborators: Nutrition 21, Inc. (Industry)
Responsible Party: Principal Investigator, Thomas L. Schwartz, M.D., Assoc Professor, State University of New York - Upstate Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: crmpicc01
Record Dates: First submitted 2008-09-24; First posted 2008-09-25 (Estimated); Last update posted 2012-09-07 (Estimated); Status verified 2012-09

CONDITIONS: Weight Gain; Obesity
Keywords: weight gain; Obesity; Psychiatry; Medication; Induced
MeSH Terms: conditions — Weight Gain; Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A,1 (Experimental): chromium piccolinate 1000mg
  Interventions: Drug: chromium piccolinate
- A,2 (Placebo Comparator): matching placebo
  Interventions: Drug: placebo for chromium piccolinate

INTERVENTIONS:
Drug: chromium piccolinate — 1000mg tab
  Arms: A,1
Drug: placebo for chromium piccolinate
  Arms: A,2

SUMMARY:
A majority of patients who suffer from mental illness are treated with serotonin regulating FDA approved medications. Some of these medications also block histamine transmission, increase blood prolactin levels, induce insulin resistance, hyperlipidemia, and promote sedation. All of which lead to weight gain and obesity. Many of these drugs are generally safe and effective but do carry the risk of a long term side effect in that acute and gradual weight gain of 10-30 pounds over a few months to a year of treatment. The detrimental gain of 7% of pre-drug weight is reported with many antipsychotics, mood stabilizers and some antidepressants. This weight gain may subsequently add to medical co-morbidity ( ie diabetes, hypertension, osteoarthritis, coronary artery diseasem, hyperlipidemia… ) This therapeutic manipulation of brain serotonin functioning may be associated with abnormal increases in carbohydrate cravings, consumption and weight gain. It is possible that insulin resistance occurs as a direct effect or as an indirect effect of weight gain, particularly in patients prone to weight gain or diabetes due to genetic loading. Leptin, a chemical associated with feedback signaling that reduces appetite and adipose tissue growth may also become insensitive. These multiple insults may lead to the worst weight gain in patients taking clozapine, olanzapine, and mirtazapine.

Diet and exercise and lifestyle modification are the usual initial interventions, though being depressed, anxious, bipolar, or schizophrenic often interferes with the ability to make these changes. In fact most of the studies which look at these weight loss interventions occur in patients who are institutionalized, on restricted diets and may respond to token economy systems while on longer term inpatient unit stays. This token economy approach is not easily translated to usual outpatient or short term inpatient practice settings. In these settings, if lifestyle modification approaches fail, patients may be placed on FDA approved diet medications (sibutramine, orlistat, ionamin…) which carry significant side effect risks. Some patients are even placed on the epilepsy medications such as zonisamide or topiramate at an even greater side effect risk.

In a similar weight gain prone group, there is growing literature in the diabetes population that the use of high dose chromium improves (lowers) insulin resistance by way of increasing insulin binding to cells, receptor numbers, and insulin receptor kinase activity. Lower fasting blood glucose levels in the blood generally occurs. Some reports show a reduction in blood lipid/cholesterol levels at higher chromium dosing as well. Recently, chromium piccolinate was studied in depressed patients, especially those with atypical features (usually fatigue, weight gain, carbohydrate cravings). Although there was no change in depression symptoms overall, carbohydrate cravings improved. This paper was presented at the 2005 American Psychiatric Association Annual Meeting in Atlanta. As a foil, a few papers in non-diabetics,non-depressed healthy volunteers showed little to no effectiveness in lowering blood sugar levels. Furthermore, one investigator (JLM) has published data showing acute , clinically significant weightgain in serotonergically treated psychiatric inpatients. The authors theorize that the use of chromium may reduce carbohydrate craving, appetite and thus protect against weight gain side effects.

Given this pivotal paper in the depressed population, effectiveness data in the diabetes population and some possible metabolic ties between these two populations, the author wishes to study the effect of chromium piccolinate in mentally ill subjects who are being started on serotonergic manipulating medications while in an inpatient treatment setting. These patients will be followed during their inpatient stay and then be followed after discharge for a single visit to determine acute interventional effects of chromium piccolinate. We feel chromium piccolinate is less toxic/hazardous than many of the weght loss medications that we currently use and therefore suggest a long term randomized, controlled study where subjects will receive active drug (chromium piccolinate) or placebo at the start of any serotonergic treatment while inpatient. The chromium piccolinate and the placbo will be obtained from the Nutrition 21 company, which has been approved by the FDA as a source of this product.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent is obtained.
* The subject is English-speaking and 18 through 64 years of age inclusive.
* The subject is currently receiving a serotonergic agent or is scheduled to receive a new or change in serotonergic psychotropic agents for their a psychiatric condition or can document that they have been on a stable regimen without any weight gain in last 3 months as a result.
* The subject must have capacity to obtain and give informed consent
* The subject must express concern about weight gain as a potential serotonin side effect.
* The patient is in good health as determined by a medical and psychiatric history, medical examination, and cannot have major medical illness that would jeopardize patient health during the study.
* Women must be of nonchildbearing potential [i.e., postmenopausal, be surgically sterile (hysterectomy or tubal ligation)] or must meet all of the following conditions: using a reliable, medically accepted form of contraception for at least 60 days before the baseline visit, and agree to continue such use throughout the duration of the study and for 30 days after the final dose of study drug. Reliable forms of contraception include oral, implanted, or injected contraceptives; intrauterine devices in place for at least 3 months; and adequate double-barrier methods in conjunction with spermicide (abstinence is considered an acceptable contraceptive regimen).
* Women must be given a urine pregnancy test (ßHCG), unless they are at least 2 years postmenopausal or surgically sterile, and the results of the test must be negative.
* The patient must be willing and able to comply with study restrictions and to remain at the clinic for the required duration during the study period, and willing to return to the clinic for the follow-up evaluation as specified in this protocol.
* The patient must be a voluntary admission inpatient at SUNY Upstate Medical University's Psychiatric department in order to enroll in the study.

Exclusion Criteria:

* The patient lacks capacity to make medical decisions and ability to receive and utilize the informed consent process due to their mental illness.
* The patient is incapacitated by mental illness
* The patient is a significant risk of suicide as determined by the study team in this acute setting
* The patient has recently started a weight loss or exercise program or is taking an insulin resistance improving drug OR plans to start one upon discharge
* The patient has a co-morbid medical problem thought to induce weight gain or make it difficult to lose weight (ie hypothyroid, hypercortisol, diabetes…)
* The patient has previously ( in the last 2 months) lost or gained a significant amount of weight from any weight loss program, weight loss agent, or dietary medication.
* The patient has used an investigational drug within 1 month before the screening visit or is participating in a concurrent clinical trial.
* The patient has any disorder that may interfere with drug absorption, distribution, metabolism, or excretion (including gastrointestinal surgery).
* The patient is highly unlikely to comply with the study protocol, be unreliable in providing ratings, or is unsuitable for any reason, as judged by the investigator.
* The patient has a clinically significant deviation from normal in the physical examination or medical history (renal or hepatic problems) which makes subject medically unstable at time of screening.
* The subject can not be currently on any medication that is clearly being used to lower weight. Examples include: Xenical, Metformin, Wellbutrin, Topomax, psycho-stimulants, and Moban.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2008-09; Primary Completion 2012-06 (Actual); Study Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
Body Weight | 6 weeks

SECONDARY OUTCOMES:
BMI | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Thomas L Schwartz, MD, Principal Investigator — SUNY Upstate; James Megna, MD, Principal Investigator — SUNY Upstate